CLINICAL TRIAL: NCT03000010
Title: Incisional Vacuum-assisted Closure Therapy After Posterior Spinal Fusion for Pediatric Neuromuscular Scoliosis
Brief Title: Wound Vac Bandage Comparison After Spinal Fusion
Acronym: WV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, G Ying Li, MD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00064814
Record Dates: First submitted 2016-12-18; First posted 2016-12-21 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Neuromuscular Scoliosis
Keywords: Wound Vac; Neuromuscular Scoliosis; Posterior Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Incisional Wound Vac (Active Comparator): We will attach sponges and a suction tube to the incision after surgery. We will leave it on for 72 hours. From then on, patients will get the care that patients normally get after spinal fusion surgery.
  Interventions: Device: Incisional Wound Vac
- Normal Gauze Bandage Group (Active Comparator): We will cover patients incision with regular gauze bandages. These are the bandages that patients normally get after spinal fusion surgery. They will be left on for 72 hours.
  Interventions: Other: Standard Bandage

INTERVENTIONS:
Device: Incisional Wound Vac
  Other Names: Incisional vacuum-assisted closure therapy
  Arms: Incisional Wound Vac
Other: Standard Bandage
  Other Names: Gauze Bandage; Gauze
  Arms: Normal Gauze Bandage Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of incisional vacuum-assisted closure (VAC) therapy in the prevention of infection after posterior spinal fusion for pediatric neuromuscular scoliosis, in comparison to a regular gauze bandage.

DETAILED DESCRIPTION:
A prospective randomized controlled study: Patients undergoing posterior spinal fusion will be randomized to a standard postoperative dressing versus an incisional VAC dressing. Both groups will have hematocrit, total lymphocyte count, and albumin checked preoperatively to assess nutritional status, drawn at the same time as standard preoperative labs during history and physical visit. Both groups will undergo standard wound closure and dressing application before breaking the sterile field. The incisional VAC group will undergo placement of an Adaptic dressing over the incision. A standard VAC sponge will be placed and secured with adhesive dressing, and a suction tube will be connected to a VAC machine set to 75 mmHg of continuous suction. The incisional VAC will be left in place for 72 hours postoperatively. Remainder of postoperative care will follow our standard posterior spinal fusion protocol and will be identical in both groups. Patients will be followed for a minimum of 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* any patient 17 years and younger
* neuromuscular scoliosis undergoing posterior spinal fusion

Exclusion Criteria:

* idiopathic and congenital scoliosis
* any type of spine surgery other than posterior spinal fusion (eg. vertical expandable prosthetic titanium rib placement, growing rod placement, anterior spinal fusion)
* intraoperative dural tear
* documented allergy to adhesive dressings

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying G Li, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Incisional Wound Vac: We will attach sponges and a suction tube to the incision after surgery. We will leave it on for 72 hours. From then on, patients will get the care that patients normally get after spinal fusion surgery.
  Incisional Wound Vac
- Normal Gauze Bandage Group: We will cover patients incision with regular gauze bandages. These are the bandages that patients normally get after spinal fusion surgery. They will be left on for 72 hours.
  Standard Bandage
Period: Overall Study
Arm/Group | Incisional Wound Vac | Normal Gauze Bandage Group
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incisional Wound Vac | Normal Gauze Bandage Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (1.6) | 12.6 (2.7) | 13 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 16 | 11 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Dehiscence or Infection
Description: Participants with wound dehiscence or infection requiring unplanned dressing changes, antibiotics, or surgery
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Incisional Wound Vac | Normal Gauze Bandage Group
Number analyzed (Participants) | 21 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data was not collected.
Description: While adverse events data was not collected, the study team discovered deaths at the time of follow-up interactions with participants' parents.
Arm/Group | Incisional Wound Vac | Normal Gauze Bandage Group
All-Cause Mortality (participants affected / at risk) | 2/21 | 2/20
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT03000010/Prot_000.pdf